CLINICAL TRIAL: NCT02730104
Title: Prospective Observational Study in Patients With Locally Advanced or Metastatic Gastroenteropancreatic Neuroendocrine Tumors Treated With Lanreotide Depot in a US Community Oncology Setting
Brief Title: Community-based Neuroendocrine Tumor (NET) Research Study
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-US-52030-340
Record Dates: First submitted 2016-04-01; First posted 2016-04-06 (Estimated); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Gastroenteropancreatic Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Cohort A: Patients with small bowel NET: Patients with small bowel NET (including appendiceal NETs)
- Cohort B: Patients with gastric NET: Patients with gastric NET (gastroduodenal)
- Cohort C: Patients with pancreatic NET
- Cohort D: Patients with colorectal NET: Patients with colorectal NET (this includes mid-gut)
- Cohort E: Unknown primary tumor

SUMMARY:
The purpose of this trial is to assess time to disease progression of patients with locally advanced or metastatic gastroenteropancreatic neuroendocrine tumors treated with Lanreotide Depot. This is an observational study therefore all data collected will be in accordance with the routine practice of physicians.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally advanced or metastatic, well-differentiated neuroendocrine tumor (NET) of the small bowel, stomach, colon/rectum, or pancreas (low or intermediate grade; i.e. G1 or G2)
* Treatment with lanreotide depot (Somatostatin Analogue-naïve patients and patients with prior treatment with octreotide long-acting repeatable (LAR) are permitted)
* Radiographically measurable disease
* Has signed the most recent written Patient Informed Consent Form

Exclusion Criteria:

* Known hypersensitivity to lanreotide
* Poorly differentiated or high grade carcinoma, or patients with neuroendocrine tumors not of lung or thymic origin
* Patients who have previously initiated treatment with lanreotide depot prior to the start of the study cannot have progressed between lanreotide initiation and study entry
* Significant history of uncontrolled cardiac disease (ie, myocardial infarction within 6 months prior to enrollment or has congestive heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-11-23; Primary Completion 2020-05-13 (Actual); Study Completion 2020-05-13 (Actual)

PRIMARY OUTCOMES:
Time to disease progression | From first date of lanreotide to up to 24 months (approximately) after the last patient is randomised
  Time to disease progression will be defined as the time from the first date of lanreotide, which may have occurred prior to study entry, to the date of first documented disease progression or the date of tumor-related death. In a living patient with no documented disease progression, or if the patient is lost to follow-up, disease progression will be censored at the date of the last evaluable scan. Patients who start a new treatment before they progress will be censored as of the date of last scan. Disease progression is defined for this study as both clinical dimensions of progression in conjunction with a treatment change.

SECONDARY OUTCOMES:
Overall survival | From first date of lanreotide to up to 24 months (approximately) after the last patient is randomised
  Overall survival will be defined as the time from the first date of lanreotide, which may have occurred prior to study entry, to the date of death due to any cause or the last date the patient was known to be alive.
Adverse events | Duration of the study, up to 24 months
Change in flushing and diarrhea | Baseline, month 6, 12, 18, 24, end of treatment visit (+/-28 days from patients off treatment)
  To be assessed as present or not, and if present, as mild, moderate, or severe. At subsequent visits, it should be noted whether these symptoms are better, worse, or the same as at previous visit.
Patient satisfaction with treatment | Month 6, 12, 18, 24, end of treatment visit (+/-28 days from patients off treatment)
  Treatment Satisfaction Questionnaire for Medication (TQSM-9)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (12):
- United States (12):
  - Arizona Oncology Associates, Sedona, Arizona
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - Texas Oncology - Beaumont, Mamie McFaddin Ward Cancer Center, Beaumont, Texas
  - Texas Oncology - Dallas Presbyterian Hospital, Dallas, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology - Denton South, Denton, Texas
  - Texas Oncology, Houston, Texas
  - Texas Oncology-Tyler, Tyler, Texas
  - Texas Oncology - Deke Slayton Cancer Center, Webster, Texas
  - Yakima Valley Memorial Hospital/North Star Lodge, Yakima, Washington

REFERENCES:
- [Derived] Paulson S, Ray D, Aranha S, Scales A, Wang Y, Liu E. Lanreotide Depot to Treat Gastroenteropancreatic Neuroendocrine Tumors in a US Community Oncology Setting: A Prospective, Observational Study. Oncol Ther. 2022 Dec;10(2):463-479. doi: 10.1007/s40487-022-00208-1. Epub 2022 Sep 22. PMID 36136274